CLINICAL TRIAL: NCT01309113
Title: Double-blind Comparison of VAC BNO 1095 Film Coated Tablets With Placebo to Identify Dose Dependent Effects in Patients Suffering From Cyclic Mastodynia and Premenstrual Syndrome
Brief Title: Dose-dependent Effects of VAC BNO 1095 on Cyclic Mastodynia and Premenstrual Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-AG-E-3
Record Dates: First submitted 2011-02-23; First posted 2011-03-04 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Cyclic Mastodynia; Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo of VAC BNO 1095 (Placebo Comparator): 1 tablet of placebo in the morning, 1 tablet of placebo in the evening
  Interventions: Drug: VAC BNO 1095 film coated tablets
- 10 mg VAC BNO 1095 (Active Comparator): 1 tablet of VAC BNO 1095 10 mg in the morning, 1 tablet of placebo in the evening
  Interventions: Drug: VAC BNO 1095 film coated tablets
- 20 mg VAC BNO 1095 (Active Comparator): 1 tablet of VAC BNO 1095 10 mg in the morning, 1 tablet of VAC BNO 1095 10 mg in the evening
  Interventions: Drug: VAC BNO 1095 film coated tablets

INTERVENTIONS:
Drug: VAC BNO 1095 film coated tablets — 3 dosages: Placebo, 10 mg of VAC BNO 1095 once daily in the morning, 10 mg of VAC BNO 1095 twice daily in the morning and in the evening

SUMMARY:
Prospective, double-blind, placebo-controlled, 3 parallel groups, multi-center study in 180 patients with cyclic mastodynia with premenstrual syndrome. 225 patients will be screened to achieve 180 patients eligible for randomisation, 60 to each treatment group, of which 150 are expected to complete the study per protocol.

Study objectives:

Identification of the optimal dosage of VAC BNO 1095 (product name) film coated tablets for treatment of cyclic mastodynia and premenstrual syndrome.

To prove the efficacy of VAC BNO 1095 film coated tablets in the treatment of cyclic mastodynia.

Dose regimen:

Group 1: VAC BNO 1095 1x10 mg:

1 tablet of verum in the morning, 1 placebo tablet in the evening

Group 2: VAC BNO 1095 2x10 mg:

1 tablet of verum in the morning, 1 tablet of verum in the evening

Group 3: Placebo:

1 tablet placebo in the morning, 1 tablet placebo in the evening

The study consists of a 2-cycle run-in period, followed by 3 cycles of treatment. After first screening further visits are scheduled after the end of each of the first and second run-in cycle, and after the first, second and third treatment cycle, respectively.

Visits will be performed during the menses at day 3 (-1+3 days), i.e. 2 days after day 1 of menstruation number n, with exception of the first screening visit which can be performed at any time prior to the first run-in cycle. Subsequently the time between the first study visit and the onset of the first run-in cycle menses T shall be added to the overall study duration.

In case that the next menstruation does not commence as expected, the patient should contact her investigator immediately in order to schedule a new appointment, approximately on the actual day 3 of the menses.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 45 who have signed an Informed Consent Form (ICF) at screening visit S-2 (screening visit -2) at the latest.
* Subject has a history of cyclic mastodynia and premenstrual syndrome
* Stable cycle duration of 25 to 35 days during the past 6 months before screening visit S-2.
* At screening visit S-2 subject is reporting at least one physical premenstrual syndrome symptom rated moderate or severe (lead symptom requiring treatment) and one psychic symptom for the late luteal phase of the preceding cycle, using the Calendar of Pre-menstrual Experiences (COPE) symptom list
* At screening visit S-2 subject is reporting symptoms of a total score of at least 15 in the late luteal phase of the preceding cycle, using the Calendar of Pre-menstrual Experiences (COPE) symptom list
* In both run-in cycles:

  * Visual analog scale greater or equal 50 mm at least on one of the days of the late luteal phase
  * Cyclic course of the mastodynia, i.e. visual analog scale in the mid follicular phase (maximum value of 5 daily recordings) is less than 75 % of the visual analog scale in the late luteal phase (maximum value of 5 daily recordings)
  * Premenstrual syndrome sum score resulting from Calendar of Pre-menstrual Experiences (COPE) must be 20 or more in the late luteal phase (average of daily recordings documented on days -5 to -1)
  * At least one physical premenstrual syndrome symptom must have been rated moderate or severe on at least one day of the late luteal phase, and one psychic symptom is present
  * Premenstrual syndrome sum score resulting from Calendar of Pre-menstrual Experiences (COPE) must not exceed 10 at day 4 of the menstruation
  * Premenstrual syndrome sum score resulting from Calendar of Pre-menstrual Experiences (COPE) must not exceed 8 in the mid follicular phase (average of daily recordings documented on days 6 to 10)

Note: "Late luteal phase" is defined as days -5 to -1 (5 days prior to the onset of menses) while "mid follicular phase" is defined as days 6 to 10 after the onset of menses.

Exclusion criteria:

* Pre- Menstrual Dysphoric Disorder
* Intake of any of the following medications before treatment start (visit S-2 up to visit V0) and within 6 months prior to visit S-2:

  * Any treatment for mastodynia or premenstrual complaints
  * Sexual hormones, combinations and inhibitors
  * Pituitary hormones and their inhibitors
  * Hypothalamic hormones
  * Neuroleptics, antidepressants
  * Serotonin-re-uptake-inhibitors
  * Prolactin-inhibitors or prolactin stimulating preparations
  * Non Steroidal Anti-Inflammatory Drugs (NSAIDs) or any other analgetics including antirheumatics
  * Spironolactone
  * Androgens
  * Gonadotrophin inhibitors
  * Diuretics
  * Danazol
  * Psychotropic agents

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in maximum severity of cyclic breast pain from baseline to visit 3 evaluated by visual analog scales | Daily from the first day of first menstruation to the last study visit (22 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Raus, MD, Study Chair — PHAMOS Central and Eastern Europe
Locations (1):
- Gynekologicko-porodnická ambulance, Olomouc, Czechia